CLINICAL TRIAL: NCT01037946
Title: Family to Family: Psychoeducation to Improve Children's Outcomes in HIV+ Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Li Li, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01NR009922 (NIH)
Record Dates: First submitted 2009-12-22; First posted 2009-12-23 (Estimated); Last update posted 2012-02-24 (Estimated); Status verified 2009-06

CONDITIONS: Quality of Life; Family Relations; Mental Health; Physical Health
Keywords: HIV; Family interventions; Thailand
MeSH Terms: conditions — Psychological Well-Being | interventions — Methods; Seroconversion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care Arm (No Intervention): Families living with HIV, offered intervention at the end of study (24 months after recruitment)
- Intervention (Experimental): Behavioral: Cognitive-behavioral, small group format sessions delivered in Thai to People Living with HIV and their caregivers once a week for 13 weeks (n=13 sessions).
  Interventions: Behavioral: Cognitive behavioral sessions

INTERVENTIONS:
Behavioral: Cognitive behavioral sessions — Behavioral: Cognitive-behavioral, small group format sessions delivered in Thai to People Living with HIV and their caregivers once a week for 13 weeks (n=13 sessions).
  Other Names: Intervention, families living with HIV
  Arms: Intervention

SUMMARY:
This project aims to support adults in HIV-affected families in order to improve their well-being. UCLA's Center for Community Health (CCH), in collaboration with the Thai Ministry of Public Health, Bureau of Epidemiology, will implement the Family-to-Family (F2F) intervention in order to improve the social, behavioral and mental health outcomes for families affected by HIV.

In Phase 1, the investigators pilot tested the current intervention contents and activities by collecting qualitative data from HIV+ families in the four district hospitals in Chiang Rai and Nakohn Ratchasima provinces selected for the proposed study. The findings from Phase was used to develop intervention content, as well as the format and style of the intervention for Phase 2. In addition, the findings from Phase 1 was used to finalize the assessment measures the investigators will use in Phase 2.

In Phase 2, 410 families with HIV+ parents from 4 district hospitals in Chiang Rai & Nakhon Ratchasima Provinces will be recruited to an intervention to benefit their school-aged children aged 6-17 years. At their clinical care site,the investigators randomly assigned families to either: 1) F2F, a psychoeducational intervention for HIV+ parents and family caregivers; or 2) a Standard Care condition. The impact of the F2F intervention will be monitored over 24 months.

DETAILED DESCRIPTION:
HIV has a negative intergenerational impact on families, particularly children with HIV+ parents. In order to improve the social, behavioral and mental health outcomes for families affected by HIV, we have designed the Family-to-Family (F2F) intervention that includes the critical, universal, program components identified by the NIMH Intervention Workgroup. All efficacious intervention programs: frame the problem by providing information and shaping beliefs; enhance skills; establish supportive relationships; and remove environmental barriers to behavior change (e.g., HIV testing, ARV). We aim to evaluate a generic intervention approach including these components that is culturally-tailored to families affected by HIV in a specific country, Thailand.

Families in Thailand need such an intervention: 1 in 4 elderly adults in Thailand will raise an AIDS orphan, even with a relatively low national seroprevalence rate (1.2%, I million adults). Thailand has a rising seroincidence. This research will design and evaluate an intervention for improving the long-term adjustment of families with HIV. We will intervene with HIV+ parents and family caregivers to improve the outcomes for families living with HIV.

The Specific Aims for the proposed study are:

1. To compare the outcomes over time of the school-age children of families in the intervention and SC conditions in each of the following domains: a) mental health symptoms; b) behavioral adjustment, and c) relationships with HIV+ parents, caregivers, and peers.
2. As intermediate outcomes, to compare the outcomes over time of the HIV+ parent in the intervention and the SC condition in terms of: health status; HIV transmission acts; parenting behaviors and bonds with children; and mental health symptoms.
3. As intermediate outcomes, to compare the outcomes over time of the partners and caregivers (about 80% grandparents) in the intervention and the SC condition in terms of: health status; mental health symptoms; caregiver burden; relationships with their HIV+ adult children, their school-age grandchildren, and bonds.
4. To compare the intermediate outcomes among those in the intervention and SC condition on disclosure and stigma-related stress.
5. To compare the influence of background factors on the impact of the intervention over time: age and gender of the HIV+ parent, the school-age child's age and gender, physical proximity in the living situation of the HIV+ parents and family caregivers, mode of initial transmission for acquisition of HIV (IDU, sexual acts), income and initial quality of relationships.

ELIGIBILITY:
Inclusion Criteria:

* HIV+ or family member of HIV+ person
* living with one or more school-age children aged 12-17;
* Informed consent;
* Disclosure of serostatus to at least one family member

Exclusion Criteria:

* No school-age children living at home; or
* No disclosure of the serostatus to any family member; or
* Inability to give informed consent or refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1033 (Actual)
Dates: Start 2005-09; Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Quality of life | Assessed up to 24 months

SECONDARY OUTCOMES:
Family relations | Assessed up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Li Li, Ph.D., Principal Investigator — University of California, Los Angeles; Sam Guo, MBA, Study Director — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States